CLINICAL TRIAL: NCT03664453
Title: A Phase 1, Open-Label, Food Effect, And Dose Proportionality Study With Omaveloxolone In Healthy Volunteers
Brief Title: A Pharmacokinetic Study of Omaveloxolone in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 408-C-1703
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: omaveloxolone; omaveloxolone capsules; RTA 408
MeSH Terms: interventions — omaveloxolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Food Effect (Fasted) (Experimental): Subjects will be randomly assigned to one of the two treatment sequences. Two single doses of omaveloxolone 150 mg (taken in multiple 50 mg capsules) will be administered to the subjects beginning in the fasted state (Period 1) with a crossover and then in the fed state (Period 2).
  Subjects will be confined beginning on Study Day -1 through the last PK blood draw on Study Day 6 during Period 1, and from Study Day 14 through the last PK blood draw on Study Day 20 during Period 2.
  Interventions: Drug: omaveloxolone
- Effect (Fed) (Experimental): Subjects will be randomly assigned to one of the two treatment sequences. Two single doses of omaveloxolone 150 mg (taken in multiple 50 mg capsules) will be administered to the subjects beginning in the fed state (Period 1) with a crossover and then in the fasted state (Period 2).
  Subjects will be confined beginning on Study Day -1 through the last PK blood draw on Study Day 6 during Period 1, and from Study Day 14 through the last PK blood draw on Study Day 20 during Period 2.
  Interventions: Drug: omaveloxolone
- Dose Proportionality (Experimental): Subjects will be randomly assigned to one of two omaveloxolone dosages. A single dose of omaveloxolone (in either 50 mg or 100 mg) will be administered to the subjects in 50 mg capsules in a fasted state.
  Subjects will be confined beginning on Study Day -1 through the last blood sample collection on Study Day 6.
  Interventions: Drug: omaveloxolone

INTERVENTIONS:
Drug: omaveloxolone — Omaveloxolone 50 mg capsules
  Other Names: RTA 408

SUMMARY:
This study will determine the effect of food on the pharmacokinetics of omaveloxolone (150 mg) in healthy adult subjects and will assess the safety, tolerability, and dose proportionality of 50 mg, 100 mg, and 150 mg omaveloxolone in healthy adult subjects.

The study will be conducted in two parts, conducted simultaneously. Part 1 will assess the food effect, while Part 2 will assess dose proportionality.

ELIGIBILITY:
Inclusion Criteria:

* Male or female and age is between 18 and 55 years, inclusive;
* All female subjects must have negative results for pregnancy tests performed;
* If male, subject must be surgically sterile or practicing at least 1 of the following methods of contraception, from initial study drug administration through 90 days after administration of the last dose of study drug;
* If male, subject agrees to abstain from sperm donation through 90 days after administration of the last dose of study drug;
* Body Mass Index (BMI) is ≥ 18 to ≤ 31 kg/m2, inclusive;
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile, and a 12-lead electrocardiogram (ECG), as judged by the investigator.

Exclusion Criteria:

* Presence or history of any significant cardiovascular, gastrointestinal, hepatic, renal, pulmonary, hematologic, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease, as determined by the investigator;
* Presence of any other condition (including surgery) known to interfere with the absorption, distribution, metabolism, or excretion of medicines;
* Requirement for any over-the-counter and/or prescription medication, vitamins, and/or herbal supplements on a regular basis;
* Recent (6-month) history of drug or alcohol abuse;
* Receipt of any investigational product within a time period equal to 10 half-lives of the product, if known, or a minimum of 30 days prior to study drug administration;
* Positive screen results for drugs of abuse, alcohol, or cotinine at screening or Day -1;
* Consumption of alcohol within 72 hours prior to study drug administration;
* Consumption of grapefruit, grapefruit products, star fruit, star fruit products, or Seville oranges within the 72-hour period prior to study drug administration;
* Use of tobacco or nicotine-containing products within the 6-month period preceding study drug administration;
* 17.10. Current enrollment in another clinical study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
Determine the effect of food on the pharmacokinetics of omaveloxolone in healthy adult subjects by measuring maximum observed concentration (Cmax) | 20 days
  Pharmacokinetics will be assessed by blood sampling for omaveloxolone to determine maximum observed concentration (Cmax).
Determine the effect of food on the pharmacokinetics of omaveloxolone in healthy adult subjects by measuring area under curve (AUC) | 20 days
  Pharmacokinetics will be assessed by blood sampling for omaveloxolone to determine area under curve (AUC).

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events | 6 days
  Safety will be assessed based on the number of treatment-emergent adverse events as defined by the Medical Dictionary for Regulatory Activities (MedDRA)

CONTACTS AND LOCATIONS:
Locations (1):
- Medpace Clinical Pharmacology Unit, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/